CLINICAL TRIAL: NCT00743964
Title: A Randomized Phase II Study of Combination Chemotherapy With Epirubicin , Cisplatin and Capecitabine (ECX) or Cisplatin and Capecitabine (CX) in Advanced Gastric Cancer
Brief Title: Phase II Study of Epirubicin, Cisplatin and Capecitabine (ECX) Versus Cisplatin and Capecitabine (CX) for Advanced Gastric Cancer (AGC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Se Hoon Park, MD, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC IRB 2008-04-027; 01-9-0804027
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Advanced Gastric Cancer
MeSH Terms: interventions — Epirubicin; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ECX (Experimental): Epirubicin, cisplatin and capecitabine combination chemotherapy will be administered.
  Interventions: Drug: Epirubicin; Drug: Cisplatin, capecitabine
- CX (Active Comparator): Cisplatin and capecitabine combination chemotherapy will be administered.
  Interventions: Drug: Cisplatin, capecitabine

INTERVENTIONS:
Drug: Epirubicin — Epirubicin 50 mg/m2 iv on day 1
  Arms: ECX
Drug: Cisplatin, capecitabine — Cisplatin 70 mg/m2 IV on day 1 of each 21 day cycle. Capecitabine 2000 mg/m2 on days 1 to 14.

SUMMARY:
Recently, 3-drug (ECX) and 2-drug (CX) combination chemotherapy involving capecitabine showed promising results in randomized clinical trials for advanced gastric cancer (AGC). The objective of the study is to evaluate the safety and activity of ECX and CX combination chemotherapy given as first-line therapy for AGC.

ELIGIBILITY:
Inclusion Criteria:

* Aged 75 years or less
* Adenocarcinoma of stomach
* Advanced, metastatic, or recurrent
* No prio chemotherapy for advanced disease
* Adequate performance status
* Adequate major organ functions

Exclusion Criteria:

* Severe comorbid illness or active infections
* Pregnancy or lactating women
* GI obstruction or malabsorption syndrome

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2008-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Failure-free survival | six months

SECONDARY OUTCOMES:
progression-free survival | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Yun J, Lee J, Park SH, Park JO, Park YS, Lim HY, Kang WK. A randomised phase II study of combination chemotherapy with epirubicin, cisplatin and capecitabine (ECX) or cisplatin and capecitabine (CX) in advanced gastric cancer. Eur J Cancer. 2010 Mar;46(5):885-91. doi: 10.1016/j.ejca.2009.12.015. Epub 2010 Jan 7. PMID 20060288